CLINICAL TRIAL: NCT03192345
Title: A Phase 1/1b First-in-human Dose Escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of SAR439459 Administered Intravenously as Monotherapy and in Combination With Cemiplimab in Adult Patients With Advanced Solid Tumors
Brief Title: A First-in-human Study of the Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of SAR439459 Monotherapy and Combination of SAR439459 and Cemiplimab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCD14678; TCD14678 (Other: Sanofi Identifier); U1111-1187-5425 (Registry Identifier: ICTRP); 2018-001113-32 (EudraCT Number)
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Malignant Solid Tumor
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Escalation monotherapy and escalation combination followed by expansion monotherapy and expansion combination. Escalation phases will not be randomized while expansion phases will be randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation SAR439459 monotherapy (Experimental): SAR439459 administered intravenously every 2 weeks in a 14-day cycle with escalating doses
  Interventions: Biological: SAR439459
- Dose Expansion SAR439459 monotherapy (Experimental): SAR439459 administered intravenously every 3 weeks in a 21-day cycle with the previously determined recommended doses as the patients will be randomized to 2 different doses
  Interventions: Biological: SAR439459
- Dose Escalation SAR439459 + cemiplimab combination (Experimental): SAR439459 + cemiplimab combination administered intravenously every 2 weeks in a 14-day cycle or every 3 weeks in a 21-day cycle with escalating SAR439459 doses and cemiplimab
  Interventions: Biological: SAR439459; Drug: Cemiplimab REGN2810
- Dose Expansion SAR439459 + cemiplimab combination (Experimental): SAR439459 + cemiplimab combination administered intravenously every 3 weeks in a 21-day cycle with previously determined SAR439459 doses and cemiplimab
  Interventions: Biological: SAR439459; Drug: Cemiplimab REGN2810

INTERVENTIONS:
Biological: SAR439459 — Pharmaceutical form: powder for solution for infusion
  Route of administration: intravenous infusion
Drug: Cemiplimab REGN2810 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous infusion
  Arms: Dose Escalation SAR439459 + cemiplimab combination; Dose Expansion SAR439459 + cemiplimab combination

SUMMARY:
Primary Objectives:

Dose escalation (Part 1)

Part 1A (SAR439459 monotherapy)

* To determine the maximum tolerated dose (MTD) and/or maximum administered dose (MAD) of SAR439459 when administered intravenously as monotherapy in adult patients with advanced solid tumors.

Part 1B (SAR439459 and cemiplimab combination therapy)

* To determine the MTD and/or MAD of SAR439459 administered intravenously in combination with cemiplimab administered intravenously in adult patients with advanced solid tumors.

Dose expansion (Part 2)

Part 2A (SAR439459 monotherapy)

* To determine optimal dose of SAR439459 administered intravenously in adult patients with advanced melanoma who have failed a prior therapy based on anti-PD-1 (programmed cell death-1) or anti-PD-L1.

Part 2B (SAR439459 and cemiplimab combination therapy)

* To determine the objective response rate (ORR) of SAR439459 in combination with cemiplimab in adult patients with selected advanced solid tumors by evaluation of antitumor response according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1).

Secondary Objectives:

* Pharmacokinetic (PK) profile SAR439459 monotherapy and combined with cemiplimab, PK profile of cemiplimab combined with SAR439459.
* Immunogenicity of SAR439459 monotherapy and combined with cemiplimab.

Dose escalation (Part 1)

* Overall safety/tolerability profile of SAR439459 monotherapy and combined with cemiplimab.
* Preliminary recommended phase 2 dose (pRP2D) of SAR439459 as monotherapy or combined with cemiplimab.

Dose expansion (Part 2)

* Progression free survival (PFS), time to progression (TTP), ORR, and safety of SAR439459 as monotherapy and PFS, TTP, duration of response (DOR), disease control rate (DCR) and safety in combination with cemiplimab.
* To confirm the optimal dose of SAR439459 administered in combination with cemiplimab.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will start from the signature of the main informed consent and include a screening period of up to 4 weeks (28 days), a treatment period of at least 1 or 2 cycles (21 or 14 days per cycle, respectively), an end-of-treatment visit at least 30 days following the last administration of study drug (or until the patient receives another anticancer therapy, whichever is earlier), and a follow-up visit 3 months after treatment discontinuation and every 3 months following, until disease progression, or initiation of another antitumor treatment, or death, whichever is earlier. For the urothelial cancer cohort in Part 2B, follow-up visits will occur every 3 months until death, study cut-off date, or upon cancellation of Survival follow-up at the discretion of the Sponsor at any prior timepoint. For the overall survival analysis (approximately 12 months after last patient first dose), whichever comes first.

Patients who have no disease progression, and continue to benefit from the study drug(s), will be allowed to continue treatment beyond the common study end-date at their assigned dose unless the study is terminated by the Sponsor. The expected enrollment period is approximately 42 months.

ELIGIBILITY:
Inclusion criteria:

Dose escalation (Part 1A and Part 1B)

* Patients with histologically confirmed, advanced unresectable or metastatic solid tumor whom in the opinion of the Investigator does not have a suitable alternative therapy.

Dose expansion (Part 2A)

* Patients with histologically confirmed, advanced unresectable or metastatic melanoma whom in the opinion of the Investigator does not have a suitable alternative therapy.
* Patients must have failed after any prior therapy based on anti-PD-1 or anti-PD-L1 as defined by disease progression within 26 weeks of initiating anti-PD-1 or anti-PD-L1 based therapy without any evidence of a response (primary resistance to anti-PD-1 or anti-PD-L1).
* Patients must have a site of disease amenable to biopsy and be a candidate for tumor biopsy. Patients must be able and willing to provide mandatory tumor biopsies prior to and during study treatment.

Dose expansion (Part 2B)

* Patients with disease location amenable to mandatory tumor biopsy at baseline with histologically confirmed advanced unresectable or metastatic melanoma, colorectal adenocarcinoma, urothelial cancer, hepatocellular carcinoma (HCC), or non-small cell lung cancer (NSCLC).
* Melanoma patients must have failed one prior therapy based on anti-PD-1 or anti-PD-L1.
* Patients with colorectal cancer must have progressed after last line of therapy.
* Patients with urothelial cancer must have disease progression during or following platinum-containing chemotherapy or within 12 months of neoadjuvant or adjuvant treatment with platinum-containing chemotherapy. Patients must not have received >2 lines of therapy for advanced disease. Patients must not have received prior treatment with anti-PD-1 or anti-PD-L1.
* Patients with HCC must have failed after 1 prior therapy based on anti-PD-1 or anti-PD-L1.
* Patients with NSCLC must have failed during or after 1 prior therapy based on anti-PD-1 or anti-PD-L1.
* Patients with histologically confirmed, advanced unresectable or metastatic melanoma, or colorectal cancer or NSCLC whom in the opinion of the Investigator do not have a suitable alternative therapy.

Dose expansion parts 2A and 2B

* At least 1 measurable lesion by RECIST v1.1.

All cohorts

* Patient understands and has signed Informed Consent form and is willing and able to comply with the requirements of the trial.

Exclusion criteria:

* Age <18 years or < the country's legal age of majority if the legal age is more than 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status >1.
* Concurrent treatment with any other anticancer therapy (including radiotherapy or investigational agents) or participation in another clinical study.
* Washout period of less than 3 weeks to prior anticancer therapy.
* Women of reproductive potential and male subjects with female partners of childbearing potential who are not willing to avoid pregnancy by using highly effective contraceptive.
* Pregnant or breast-feeding women.
* Unwillingness and inability to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
* Significant and uncontrolled concomitant illness, including any psychiatric condition.
* Active infections, including unexplained fever (temperature >38.1ºC), or antibiotic therapy within 1 week prior to enrollment.
* Any prior organ transplant including allogeneic bone marrow transplant.
* History within the last 5 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* History of known human immunodeficiency virus (HIV), HIV serology at screening will be conducted only for patients in German study sites.
* Known uncontrolled hepatitis B virus (HBV) infection.
* Known untreated current hepatitis C virus (HCV) infection.
* Any major surgery within the last 28 days.
* Patients with primary central nervous system (CNS) tumors and/or CNS metastases of non-CNS primary tumors.
* History of congestive heart failure, myocardial infarction with reduced ejection fraction, symptomatic coronary artery disease, documented uncontrolled hypertension, major clinically significant Electrocardiography (ECG) and echocardiogram abnormalities, significant ventricular arrhythmias, significant valvular heart disease (including valve replacement), vascular malformation, aneurysm, significant pulmonary conditions such as idiopathic pulmonary hypertension, uncontrolled chronic lung disease.
* History of severe, acute or chronic renal diseases.
* Any of the following within 6 months prior to study enrollment: pulmonary embolism, deep vein thrombosis, active uncontrolled bleeding, infectious or inflammatory bowel disease, diverticulitis, intestinal obstruction or perforation and gastrointestinal hemorrhage.
* Inadequate hematological, renal or liver function.
* Non-resolution of any prior treatment related toxicity to Grade <2.
* Prior treatment with any anti-transforming growth factor β (anti-TGFβ) inhibitors.
* Known allergies to any component of SAR439459 and/or cemiplimab.
* Patients with uveal melanoma and patients with prior or ongoing uveitis.
* Patients who received prior immunotherapy who developed toxicity leading to a permanent discontinuation of immunotherapy.
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments.
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of SAR439459 and/or cemiplimab (occasional use of inhaled, intraocular, nasal or topical steroids for symptomatic relief allowed).
* History of interstitial lung disease or active non-infectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
* Patients with underlying cancer predisposition syndromes.
* Receipt of a live vaccine within 30 days of planned start of study medication.
* Therapeutic doses of anticoagulants or antiplatelet agents within 7 days prior the first dose of SAR439459.
* Prothrombin time (PT) or international normalized ratio (INR) > 1.5 × upper limit of normal (ULN).
* Patients accommodated in an institution because of regulatory or legal order; prisoners or patients who are legally institutionalized.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Through the end of 1 or 2 cycles, total duration up to 6 weeks (for Part 1A each cycle is 2 weeks; for Part 1B each cycle is 2 or 3 weeks)
  Incidence of DLTs at Cycle 1 and/or 2 in Parts 1A and 1B.
Objective Response Rate (ORR) for Part 2B | Continuous throughout study assessment (up to approximately 1 year)
  Efficacy as documented by ORR will be assessed by evaluation of antitumor response information according to RECIST 1.1 (Part 2B).

SECONDARY OUTCOMES:
Overall safety profile | Continuous throughout study assessment (up to approximately 1 year)
  The overall safety profile of SAR439459 administered in monotherapy (Part 1A and Part 2A) or in combination with cemiplimab (Part 1B and Part 2B).
Progression free survival (PFS) | Continuous throughout study assessment (up to approximately 1 year)
  The time from first investigational medicinal product (IMP) administration until objective tumor progression or death (Part 2A and Part 2B).
Time to progression (TTP) | Continuous throughout study assessment (up to approximately 1 year)
  The time from first IMP administration until objective tumor progression (Part 2A and 2B).
Objective Response Rate (ORR) Part 2A | Continuous throughout study assessment (up to approximately 1 year)
  Efficacy as documented by ORR will be assessed by evaluation of antitumor response information according to RECIST 1.1 (Part 2A).
Duration of response Part 2B | Continuous throughout study assessment (up to approximately 1 year)
  Time from initial response to the first documented tumor progression.
Disease Control Rate Part 2B | Continuous throughout study assessment (up to approximately 1 year)
  Sum of complete response, partial response and stable disease rates
Immunogenicity evaluation | Up to approximately 1 year
  Blood samples will be assessed for human anti-SAR439459 antibodies (all cohorts) and for human anti-cemiplimab antibodies (Parts 1B and 2B).
Cmax for SAR439459 and for cemiplimab | Cycle 1, Day 1 to Day 15 or to Day 22
  Maximum plasma concentration observed.
AUC for SAR439459 | Cycle 1, Day 1 to Day 15 or to Day 22
  Area under the serum concentration versus time curve extrapolated to infinity.
AUC0-tau for SAR439459 and for cemiplimab | Cycle 1, Day 1 to Day 15 or to Day 22
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to 14 or 21 days post-dose.
t1/2z for SAR439459 | Cycle 1, Day 1 to Day 15 or to Day 22
  Terminal half-life associated with the terminal slope (λz).
CL for SAR439459 | Cycle 1, Day 1 to Day 15 or to Day 22
  Total body clearance of a drug from plasma calculated using the following equation from AUC: CL= Dose/AUC on cycle 1.
Vss for SAR439459 | Cycle 1, Day 1 to Day 15 or to Day 22
  Estimate of Volume of distribution at the steady state after single intravenous dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (34):
- United States (6):
  - The University of Kansas Clinical Research Center Site Number : 8400004, Fairway, Kansas
  - Massachusetts General Hospital Site Number : 8400001, Boston, Massachusetts
  - Dana Farber Cancer Institute Site Number : 8400101, Boston, Massachusetts
  - Duke University Medical Center Site Number : 8400008, Durham, North Carolina
  - Tennessee Oncology, PLLC Site Number : 8400006, Nashville, Tennessee
  - Mary Crowley Cancer Research Center Site Number : 8400003, Dallas, Texas
- Australia (2):
  - Investigational Site Number : 0360002, Heidelberg West, Victoria
  - Investigational Site Number : 0360001, Melbourne, Victoria
- Investigational Site Number : 0560001, Leuven, Belgium
- Canada (3):
  - Investigational Site Number : 1240003, Calgary, Alberta
  - Investigational Site Number : 1240001, Toronto, Ontario
  - Investigational Site Number : 1240002, Montreal, Quebec
- Investigational Site Number : 2330001, Tallinn, Estonia
- France (4):
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500003, Nantes
  - Investigational Site Number : 2500005, Nantes
  - Investigational Site Number : 2500001, Villejuif
- Germany (2):
  - Investigational Site Number : 2760001, Essen
  - Investigational Site Number : 2760003, Hanover
- Italy (3):
  - Investigational Site Number : 3800003, Rozzano, Milano
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800002, Milan
- Netherlands (2):
  - Investigational Site Number : 5280001, Rotterdam
  - Investigational Site Number : 5280002, Utrecht
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (5):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240005, Pamplona, Navarre
- Investigational Site Number : 1580002, Tainan, Taiwan
- United Kingdom (2):
  - Investigational Site Number : 8260001, Glasgow, Central Bedfordshire
  - Investigational Site Number : 8260002, Cardiff, Vale of Glamorgan, the

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Baranda JC, Robbrecht D, Sullivan R, Doger B, Santoro A, Barve M, Grob JJ, Bechter O, Vieito M, de Miguel MJ, Schadendorf D, Johnson M, Pouzin C, Cantalloube C, Wang R, Lee J, Chen X, Demers B, Amrate A, Abbadessa G, Hodi FS. Safety, pharmacokinetics, pharmacodynamics, and antitumor activity of SAR439459, a TGFbeta inhibitor, as monotherapy and in combination with cemiplimab in patients with advanced solid tumors: Findings from a phase 1/1b study. Clin Transl Sci. 2024 Jun;17(6):e13854. doi: 10.1111/cts.13854. PMID 38898592
- [Derived] Greco R, Qu H, Qu H, Theilhaber J, Shapiro G, Gregory R, Winter C, Malkova N, Sun F, Jaworski J, Best A, Pao L, Hebert A, Levit M, Protopopov A, Pollard J, Bahjat K, Wiederschain D, Sharma S. Pan-TGFbeta inhibition by SAR439459 relieves immunosuppression and improves antitumor efficacy of PD-1 blockade. Oncoimmunology. 2020 Sep 13;9(1):1811605. doi: 10.1080/2162402X.2020.1811605. PMID 33224628